CLINICAL TRIAL: NCT00770172
Title: Moderate Persistent Neutropenia: Comparison of Administration of G-CSF (Granulocyte Colony Stimulating Factor) 1 Day Out of 2 Versus Traditional Schedules to Maintain Dose Intensity. Phase III Multicenter Study in Patients With Solid Tumors Receiving Chemotherapy
Brief Title: G-CSF in Preventing Neutropenia in Patients With Solid Tumors Who Are Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000599523; FRE-CFB-LENO-12; INCA-RECF0515; EUDRACT-2007-002742-38; CFB-2007-02; CHUGAI-FRE-CFB-LENO-12
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2008-12

CONDITIONS: Chemotherapeutic Agent Toxicity; Neutropenia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: chemotherapeutic agent toxicity; neutropenia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neutropenia | interventions — Filgrastim

ARMS (2):
- Arm I (Experimental): Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily for 6 days beginning 1 week after the start of chemotherapy (days 7-12). If chemotherapy begins on day 8, patients receive G-CSF SC on days 9-14.
  Interventions: Biological: filgrastim
- Arm II (Experimental): Patients receive G-CSF SC every 2 days on days 10-20 for up to 6 injections.
  Interventions: Biological: filgrastim

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously

SUMMARY:
RATIONALE: Colony-stimulating factors, such as G-CSF, may increase the number of white blood cells found in bone marrow or peripheral blood and may prevent persistent neutropenia in patients receiving chemotherapy. It is not yet known which regimen of G-CSF may be more effective in preventing neutropenia.

PURPOSE: This randomized phase III trial is comparing two different regimens of G-CSF to see how well it works in preventing persistent neutropenia in patients with solid tumors who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of filgrastim (G-CSF) in preventing persistent moderate neutropenia in patients with solid tumors while maintaining chemotherapy courses.

Secondary

* Compare the tolerability of 2 regimens of G-CSF in these patients.
* Determine the number of courses of G-CSF needed in each regimen.
* Evaluate the frequency of infections.
* Determine dose intensity.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily for 6 days beginning 1 week after the start of chemotherapy (days 7-12). If chemotherapy begins on day 8, patients receive G-CSF SC on days 9-14.
* Arm II: Patients receive G-CSF SC every 2 days on days 10-20 for up to 6 injections.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor
* Receiving chemotherapy in any line of treatment (adjuvant or metastatic)

  * Chemotherapy courses repeating every 21 days or beginning on day 8 allowed
  * Received at least 2 prior courses of chemotherapy
* Moderate neutropenia (grade 1-3) leading to a delay of the first course by ≥ 7 days or a delay of the second course of treatment

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known hypersensitivity to filgrastim (G-CSF) or any of its components
* No severe immunodepression
* No malignant hematological disease
* No history of psychiatric illness
* No patients deprived of liberty or under guardianship
* No psychological, familial, social, or geographical reasons preventing follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of courses of G-CSF required

CONTACTS AND LOCATIONS:
Overall Officials: Florence Joly, MD, PhD, Study Chair — Centre Francois Baclesse
Locations (1):
- Centre Regional Francois Baclesse, Caen, France